CLINICAL TRIAL: NCT05587634
Title: Virtual Peer Health Coaching as an Effective Intervention for Increasing Physical Activity in Adolescents With Physical Disability
Brief Title: Virtual Peer Health Coaching for Adolescents With Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Principal Investigator, Cheri Blauwet, Associate Professor of Physical Medicine and Rehabilitation, Harvard Medical School, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019P003354
Record Dates: First submitted 2022-09-13; First posted 2022-10-20 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy; Spina Bifida
MeSH Terms: conditions — Cerebral Palsy; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Health Coaching Intervention (Experimental): Intervention Arm - these participants receive individualized peer health coaching (intervention group only) and an adaptive physical activity guide of local resources (both groups)
  Interventions: Behavioral: Virtual Peer Health Coaching
- Control (No Intervention): Control arm - these participants receive only an adaptive physical activity local guide including information on local adaptive sports opportunities however no individualized peer health coaching

INTERVENTIONS:
Behavioral: Virtual Peer Health Coaching — Intervention arm: weekly sessions (~30 min each session) of physical activity counseling with an assigned peer health coach over the course of 12 weeks. The focus of the initial 2 calls is on rapport development and trust building with a focus around PA with discussion of physical activity goals and motives, where possible. The remainder of the call sessions follow a standardized format of a 30-minute call to 1) review the previous week, 2) integrate motivational strategies, and 3) develop action and support plans for the next week. The final call format includes a summary and evaluation of the intervention, discussion of short- and long-term goals, and relapse prevention strategies. Sessions guided by a call tracking form.
  These participants receive an adaptive physical activity local guide including information on local adaptive sports opportunities, which the control group also receives.
  Arms: Peer Health Coaching Intervention

SUMMARY:
Participation in physical activity (PA) confers clear physical and psychosocial benefits. Yet, many adolescents with physical disabilities such as cerebral palsy and spina bifida do not engage in regular PA, putting them at increased risk for the detrimental impact of sedentary lifestyles such as high rates of obesity/overweight - adverse health trends that continue into adulthood. To address this PA gap, a feasibility pilot randomized controlled trial is proposed evaluating the utility of a peer health coach intervention to promote PA participation and to improve outcomes related to self-autonomy, self-efficacy, and quality of life in adolescents with physical disabilities. Peer health coaches will themselves be young adults with disabilities, trained in concepts of motivational interviewing and self-determination theory, enabling them to meet participants "where they are at" in their understanding of PA and readiness to change PA behaviors. This study will be novel given that: 1) for the first time, an adult peer health coaching model targeting PA will be adapted to the needs of adolescents with disabilities, 2) the study will employ text messaging and other social media platforms that are highly relevant to an adolescent population, and 3) the study will assess PA participation with use of ActiGraph activity trackers, designed to monitor both duration and intensity of PA in individuals with mobility impairment. The results of this study will be used to inform the design of a future, definitive RCT evaluating the efficacy of a peer health coaching intervention to create meaningful change in physical and psychosocial outcomes. By empowering adolescents with disabilities to take control of their own physical and psychosocial health, this work has the potential to impact the well-being and quality of life of participants for many years to come.

DETAILED DESCRIPTION:
Physical activity is an often overlooked, yet incredibly powerful, tool for empowering adolescents with disabilities to take control of their own physical and psychosocial health. At least 60 minutes of daily physical activity (PA) is recommended for children and adolescents ages 6-17, yet the vast majority of young people with disabilities do not meet these goals. As a result, children and adolescents with disabilities are more likely than their non-disabled peers to experience the detrimental impact of sedentary lifestyles such as high rates of obesity/overweight - adverse health trends that continue into adulthood. Additionally, given that children and adolescents with disabilities remain systematically excluded from community and school-based sports and PA opportunities - a mainstay of social development and confidence-building in able-bodied youth - those with disabilities are more likely to experience social isolation and thus threats to well-being and quality of life.

In this context, prior research has focused on the role of peer health coaching (PHC) to enhance health self-management in individuals with disabilities, demonstrating efficacy in reducing rates of secondary conditions and improving self-efficacy and life satisfaction. PHCs simultaneously act as advisor, supporter, and role model, providing the "hook" that stimulates behavior change. Although the PHC model has also been used to promote participation in PA, studies have focused on adults primarily with spinal cord injury. While it is well known that engagement in PA in adolescence is correlated with similar behaviors in adulthood, no prior trials have explored the efficacy of PHCs in stimulating PA behavior in adolescents with childhood-onset disability.

To explore effective solutions that stimulate PA participation to promote equity and quality of life in adolescents with disabilities, this pilot study will target adolescents with cerebral palsy (CP) and spina bifida (SB), the 2 most common types of childhood-onset physical disability, with the following specific aims:

Primary Objective:

To evaluate the feasibility of conducting an efficacy trial of the first virtual PHC intervention aimed to increase PA participation in adolescents with CP and SB. This will include assessing the acceptability of the intervention to our key stakeholders - adolescents with disabilities and their families.

Secondary Objective:

To determine the responsiveness of selected outcome measures to the first virtual PHC intervention in adolescents with CP and SB. Outcomes will include the assessment of a) physical activity, b) psychosocial health, and c) quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12-17 years
* Primary residence in cities and towns within greater Boston
* Presence of CP or SB resulting in mobility limitation
* CP - Gross Motor Function Classification System (GMFCS) level II and III
* SB - myelomeningocele, lipomyelomeningocele, or tethered cord syndromes with motor impairment
* Fluent in conversational English
* Able to utilize a personal cell phone for verbal and text message communications
* Intentions of engaging in PA

Exclusion Criteria:

* Presence of significant cognitive impairment - IQ below 55 as measured by Wechsler Intelligence Score for Children (WISC) or Wechsler Adult Intelligence Scale (WAIS), or those below a 3rd grade reading level
* Use of power mobility as the primary form of mobility on a daily basis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility measure: Recruitment | Months 1-12 for the overall study
  Measuring feasibility of recruitment by measuring ability to reach goal of three to four participants/month are recruited over 12 months (for target n=40)
Feasibility measure: Recruitment | Months 1-12 for the overall study
  Measuring feasibility of recruitment by measuring ability to reach goal of >10% of eligible individuals approached for recruitment are recruited
Feasibility: Stratification for age | Months 1-12 for the overall study
  Measuring balance of recruitment by goal of intervention/control groups being balanced for age
Feasibility: Stratification for sex | Months 1-12 for the overall study
  Measuring balance of recruitment by goal of intervention/control groups being balanced for sex (male versus female)
Feasibility: Stratification for diagnosis | Months 1-12 for the overall study
  Measuring balance of recruitment by goal of intervention/control groups being balanced for diagnosis
Feasibility: Attrition | Months 1-3 for participants; Months 1-15 of overall study
  Measuring feasibility of participation by measuring ability to meet goal of having >80% of individuals complete all outcome measures
Feasibility: Participant Engagement and Adherence to Intervention with Coach | Months 1-3 for intervention participants; Months 1-15 of overall study
  Measuring feasibility of participant engagement and adherence to intervention by measuring ability of intervention group participants to complete the goal of >75% of calls with peer health coach
Feasibility: Participant Engagement and Adherence to Intervention: Post Call Questionnaires | Months 1-3 for intervention participants; Months 1-15 of overall study
  Measuring feasibility of participant engagement and adherence to intervention by measuring ability of intervention group participants to complete the goal of >75% of post call questionnaires
Feasibility: Peer Health Coach Engagement and Implementation of Intervention: Checklist | Months 1-3 for intervention participants; Months 1-15 of overall study
  Measuring feasibility of peer health coach engagement and implementation of intervention by measuring ability of Peer Health Coaches to complete the coaching intervention checklist with a goal of completion in >90% of sessions with intervention participant mentee
Feasibility: Peer Health Coach Engagement and Implementation of Intervention: Questionnaires | Months 1-3 for intervention participants; Months 1-15 of overall study
  Measuring feasibility of peer health coach engagement and implementation of intervention by ability of peer health coaches to complete a goal of >90% of post call questionnaires
Feasibility: Peer Health Coach Engagement and Implementation of Intervention: Coaching Sessions | Months 1-3 for intervention participants; Months 1-15 of overall study
  Measuring feasibility of peer health coach engagement and implementation of intervention by measuring the ability of Peer Health Coaches to complete full coaching session within 1 hour, including preparation, documenting call content, and post call questionnaires
Acceptability: Intervention Participants Qualitative Satisfaction with Peer Health Coach Intervention | Month 3 (after completion of intervention) for intervention participants
  Measuring acceptability of peer health coach intervention through qualitative analysis of data from semi-structured interview. After completion of intervention, each intervention participant has a semi-structured interview with the research team, with questions about satisfaction with peer health coach intervention.
Acceptability: Intervention Participants Quantitative Satisfaction with Peer Health Coach Intervention | Month 3 (after completion of intervention) for intervention participants
  Measuring acceptability of peer health coach intervention through a quantitative questionnaire with 3 questions that are using a scale of "No effort" to "Every Effort" regarding perceptions of the peer health coach's efforts in helping the intervention group participant meet their goals.
Acceptability: Intervention Participants Qualitative Impact of Peer Health Coach Intervention | Month 6 (3 months post-intervention) for intervention participants
  Measuring acceptability of peer health coach intervention through qualitative analysis of data from semi-structured interview. Three months after completion of intervention, each intervention participant has a semi-structured interview with the research team, with questions about ongoing impact of peer health coaching intervention on removing physical activity barriers.
Acceptability: Intervention Participants Evaluation of Collaboration of the Peer Health Coach | Month 3 (after completion of intervention) for intervention participants
  Measuring the quality of the peer health coach collaboration through survey question provided to the intervention group participants after completed of the intervention. Percentage scale used from 0% to 100% rating of the collaboration, with higher numbers indicating greater collaboration.

SECONDARY OUTCOMES:
Actigraph Electronic Physical Activity Tracker Compliance | Months 1-3 for participants; Months 1-15 of overall study
  Measuring Actigraph Electronic Physical Activity Tracker compliance by measuring if compliance reaches a goal of 80% of participants assigned to wear Actigraph physical activity tracker (e.g., 50% of intervention group and 50% of control group) wearing the Actigraph at least 5 hours daily at least 4/7 days weekly averaged over a 4-week period throughout the 3-month period
Arc Self-Determination Scale | At the following time points for participants: 6 weeks, 12 weeks, 6 months
  Self-determination will be evaluated via the Arc Self-Determination Scale (ASDS), which is reliable and valid in adolescents with disability. There are 72 questions on the Arc Self-Determination Scale and the scoring is completed by taking raw values and comparing them against a normative value chart which then indicates the percentile of the scoring rather than using the raw values alone. Higher percentiles indicate higher self determination.
The PedsQL Measurement Model for the Pediatric Quality of Life Inventory | At the following time points for participants: 6 weeks, 12 weeks, 6 months
  This is a validated scale to measure quality of life (ages 5-18) in terms of school functioning and physical, emotional and social health. This is well-researched in individuals with cerebral palsy and spina bifida. The scale is from 0 to 100, with higher scores indicating higher health-related quality of life.
Physical Activity Self-Efficacy Scale: Adolescent Protocol | At the following time points for participants: 6 weeks, 12 weeks, 6 months
  The Physical Activity Self-Efficacy Scale will test self-efficacy/confidence in physical activity engagement under challenging circumstances, and has good internal consistency and test-retest reliability. The scale is from 8 to 40 with higher scores indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri Blauwet, MD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbone PS, Smith PJ, Lewis C, LeBlanc C. Promoting the Participation of Children and Adolescents With Disabilities in Sports, Recreation, and Physical Activity. Pediatrics. 2021 Dec 1;148(6):e2021054664. doi: 10.1542/peds.2021-054664. PMID 34851421
- [Background] Houlihan BV, Brody M, Everhart-Skeels S, Pernigotti D, Burnett S, Zazula J, Green C, Hasiotis S, Belliveau T, Seetharama S, Rosenblum D, Jette A. Randomized Trial of a Peer-Led, Telephone-Based Empowerment Intervention for Persons With Chronic Spinal Cord Injury Improves Health Self-Management. Arch Phys Med Rehabil. 2017 Jun;98(6):1067-1076.e1. doi: 10.1016/j.apmr.2017.02.005. Epub 2017 Mar 8. PMID 28284835
- [Background] Houlihan BV, Everhart-Skeels S, Gutnick D, Pernigotti D, Zazula J, Brody M, Burnett S, Mercier H, Hasiotis S, Green C, Seetharama S, Belliveau T, Rosenblum D, Jette A. Empowering Adults With Chronic Spinal Cord Injury to Prevent Secondary Conditions. Arch Phys Med Rehabil. 2016 Oct;97(10):1687-1695.e5. doi: 10.1016/j.apmr.2016.04.005. Epub 2016 Apr 30. PMID 27143581
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Kleis RR, Hoch MC, Hogg-Graham R, Hoch JM. The Effectiveness of the Transtheoretical Model to Improve Physical Activity in Healthy Adults: A Systematic Review. J Phys Act Health. 2021 Jan 1;18(1):94-108. doi: 10.1123/jpah.2020-0334. Epub 2020 Dec 1. PMID 33260143
- [Background] Young MD, Plotnikoff RC, Collins CE, Callister R, Morgan PJ. Social cognitive theory and physical activity: a systematic review and meta-analysis. Obes Rev. 2014 Dec;15(12):983-95. doi: 10.1111/obr.12225. Epub 2014 Oct 7. PMID 25428600